CLINICAL TRIAL: NCT07172295
Title: Modulate Tremor Severity With Low-intensity Focused Ultrasound Stimulation Targeting the Deep Nucleus of Patients With Refractory Hand Tremor.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, National Taiwan University Hospital, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202405134DINC
Record Dates: First submitted 2025-08-11; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease (PD); Essential Tremor; Dystonic Tremor; Continuous Theta Burst Stimulation Transcranial Focused Ultrasound
Keywords: NaviFUS; Tremor; Transcranial focused ultrasound
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tremor treatment (Experimental)
  Interventions: Procedure: Accelerated NaviFUS-ctbFUS stimulation

INTERVENTIONS:
Procedure: Accelerated NaviFUS-ctbFUS stimulation — Three consecutive sessions of NaviFUS-ctbTUS stimulation were performed, with a 5-minute interval between each session.
  The acoustic pressure was set such that the estimated intracranial pressure at 30% skull transmission was approximately 0.5 MPa.
  The stimulation target was the center of the Vop, with a total of 7 stimulation points.

SUMMARY:
The study plans to recruit 12 patients with Parkinsonian tremor, essential tremor, or dystonic tremor. After receiving NaviFUS-ctbTUS stimulation, the improvement in their tremor will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years.
* Subjects must belong to one of the following three categories:

  1. Patients with Parkinson's disease tremor who have an inadequate response to medication.
  2. Patients with essential tremor who have an inadequate response to medication.
  3. Patients with dystonic tremor who have an inadequate response to medication.
* Subjects are willing to shave hair over the treatment area for focused ultrasound.
* Stable medication regimen (types and dosages) for at least 4 weeks prior to study enrollment.
* Normal liver and renal function (Creatinine < 1.3 mg/dL, GPT < 41 U/L).
* Female participants of childbearing potential, or male participants with female partners of childbearing potential, must agree to use appropriate contraception from the first study treatment until at least 6 months after the last treatment to prevent pregnancy.

Exclusion Criteria:

* Presence of intracranial implants deemed unsuitable for MRI, such as metal clips, ventriculoperitoneal (VP) shunts, cochlear implants, deep brain stimulation (DBS) devices, pacemakers, or implantable cardioverter- defibrillators (ICDs).
* Any abnormalities along the focused ultrasound beam path through the skull, including scars on the skull, scalp conditions (e.g., eczema), open wounds, calp atrophy, or significant calcification confirmed by imaging along the ultrasound transmission pathway.
* Pregnant or breastfeeding women.
* Use of investigational drugs from other clinical trials.
* Patients with major depressive disorder (Beck Depression Inventory-II score > 30 within the past year) or with suicidal ideation.
* Any condition that, in the opinion of the investigator, may interfere with treatment efficacy or increase risk to the subject.
* Presence of any brain tumors, vascular malformations, or significant traumatic brain injury.
* Presence of significant psychiatric symptoms (Clinical Dementia Rating [CDR]

  * 2).
* Use of anticoagulant medications.
* Use of medications known to exacerbate tremor.
* Tremor due to metabolic or psychogenic causes.
* Coagulopathy or abnormal coagulation profiles, including any of the following:

  1. Platelet count ≤ 100,000/µL
  2. INR ≥ 1.5
  3. PT ≥ 1.5 × upper limit of normal (ULN)
  4. aPTT ≥ 1.5 × ULN
  5. Fibrinogen ≤ 150 mg/dL
* Inability to provide informed consent or comply with study procedures, posing potential safety concerns.
* Insufficient skull density as determined by pre-treatment evaluation, resulting in ultrasound transmission efficiency less than 20%.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events Compared to Baseline [Safety Assessment] | Day of first stimulation, 7 days after first stimulation, day of second stimulation, 7 days after second stimulation, and 28 days after second stimulation.
  The safety of using the NaviFUS system in patients with tremor will be assessed throughout the study period. Any examination result that shows a significant change compared to baseline (Visit 1), as determined by the investigator, will be documented and reported as an adverse event (AE).

SECONDARY OUTCOMES:
Change in Tremor Amplitude [Efficacy] | On the day of first stimulation and the day of second stimulation: immediately before treatment, and at 0, 20, 40, and 60 minutes post-treatment; on the day of second stimulation, also after task-based fMRI.
  Efficacy will be assessed by determining whether there is a change in tremor amplitude across multiple time points following treatment. Measurements (archimedes spirogram ) will be taken pre-treatment and at several time points post-treatment to evaluate immediate and short-term effects.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch, Hsinchu, Hsinchu City, Taiwan